CLINICAL TRIAL: NCT05472467
Title: Camrelizumab Combination With SBRT and Concurrent Chemotherapy Treated Stage IV Oligometastatic Non-small Cell Lung Cancer ，a Single-arm, Single-center, Exploratory Clinical Study（IMCORT-2）
Brief Title: Camrelizumab Combination With SBRT and Concurrent Chemotherapy Treated Stage IV Oligometastatic Non-small Cell Lung Cancer
Acronym: IMCORT-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, LI TAO, Section Head, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCHEC-01-2021-091
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: NSCLC,Camrelizumab,SBRT,oligometastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; Radiosurgery; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy combined with Stereotactic Body Radiation Therapy (Experimental): 1. Camrelizumab： 200mg IV Q3W
  2. Chemotherapy：Squamous carcinoma: docetaxel 60 mg/m2, d1 + cisplatin 25 mg/m2, d1-3 or carboplatin AUC=4-6 d1, 21 days for one cycle, up to 4 cycles.
     Non-squamous carcinoma: pemetrexed 500 mg/m2, d1 + cisplatin 25 mg/m2, d1-3 or carboplatin AUC=4-6, d1,21 days for one cycle, up to 4 cycles.
  3. Stereotactic Body Radiation Therapy(SBRT) for Oligometastatic the total dose 35Gy/5f(7.0Gy/f,5f per week)。
  Interventions: Drug: Camrelizumab; Radiation: stereotactic body radiation therapy; Drug: Chemotherapy

INTERVENTIONS:
Drug: Camrelizumab — 200mg IV Q3W. Every three weeks is a cycle
Radiation: stereotactic body radiation therapy — stereotactic body radiation therapy for Oligometastases 35Gy/5f(7.0Gy/f,5f per week)
  Other Names: SBRT
Drug: Chemotherapy — Squamous carcinoma: docetaxel 60 mg/m2, d1 + cisplatin 25 mg/m2, d1-3 or carboplatin AUC=4-6 d1, 21 days for one cycle, up to 4 cycles.
  Non-squamous carcinoma: pemetrexed 500 mg/m2, d1 + cisplatin 25 mg/m2, d1-3 or carboplatin AUC=4-6, d1,21 days for one cycle, up to 4 cycles.

SUMMARY:
This study evaluated the effectiveness and safety of Camrelizumab combination with SBRT and concurrent chemotherapy treated stage IV oligometastatic non-small cell lung cancer

DETAILED DESCRIPTION:
This study evaluated the effectiveness and safety of Camrelizumab combination with SBRT and concurrent chemotherapy treated stage IV oligometastatic non-small cell lung cancer.

The primary endpoint is ORR. Secondary points contains：PFS、OS、DCR、Qol.

ELIGIBILITY:
Inclusion Criteria:

1. patients voluntarily enrolled in this study and signed the informed consent form (ICF).

   Good compliance and cooperation with follow-up.
2. age: 18 to 75 years, both sexes.
3. ECOG PS: 0 to 1 score.
4. patients with non-small cell lung cancer clearly diagnosed by pathology, with measurable tumor lesions (oligometastases ≥10 mm in length, meeting mRECIST1.1 criteria).
5. subjects with clinical stage IV according to the 8th edition of the Clinical Oncology TNM staging Stage IV (≤5 oligometastases, ≤3 metastatic organs, and measurable metastases) non-small cell lung cancer patients according to the 8th edition of TNM staging.

5. patients with stage IV clinical stage (number of oligometastases ≤ 5, metastatic organs ≤ 3, and measurable metastases) non-small cell lung cancer 6. vital organ function meets the following requirements (no blood components and cell growth are allowed 2 weeks prior to the start of study treatment) (No blood components or cell growth factors are allowed 2 weeks prior to the start of study treatment).

(1) Routine blood tests must meet the following requirements.

1. absolute neutrophil count (ANC) ≥ 1.5 x 109

   * L.
2. Hemoglobin (HB) ≥ 9 g/dL.
3. Platelets (PLT) ≥ 100×109 /L.
4. serum albumin (ALB) ≥ 2.8g/dL. (2) Biochemical examination shall comply with.

a) total bilirubin (TBIL) ≤ 1.5 ULN. b) ALT, AST ≤ 2.5 UILN (if liver function abnormalities due to liver metastases, then ≤ 5 ULN) b) ALT, AST ≤ 2.5 UILN (≤ 5 ULN if liver function abnormalities are due to liver metastasis).

c) serum creatinine sCr ≤ 1.5 ULN, endogenous creatinine clearance c) serum creatinine sCr ≤ 1.5 ULN and endogenous creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula).

7. expected survival ≥ 3 months. 8. the patient is judged by the investigator to be amenable to treatment with kallikreinumab 9. the patient has no autoimmune disease. 10. the patient has not received prior treatment with PD-1/PD-L1 inhibitors. 11. tissue or plasma genetic testing for common lung cancer driver genes such as EGFR, ALK, ROS, RET, HER2, MET, BRAF negative, or no accessible targeted drugs or who are intolerant to targeted drug therapy.

12. Female subjects of childbearing potential should receive their first study drug administration within 12. Female subjects of childbearing potential should have a urine or serum pregnancy test within 72 hours prior to the first study drug administration and demonstrate 12. Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to the first dose of study drug and be willing to use validated methods during the trial until 3 months after the last administration of cariolizumab. Male subjects whose partners are women of childbearing potential should use an effective method of contraception for the duration of the trial and for 3 months after the last administration of cariolizumab. Male subjects whose partners are women of childbearing potential should use an effective method of contraception during the trial and for 3 months after the last administration of carreliximab

Exclusion Criteria:

1. patients who do not meet the inclusion criteria for type of pathology and site of primary focus.
2. with diffuse brain metastases and meningeal metastases
3. have any active autoimmune disease or a history of autoimmune disease such as inter stromal pneumonia, uveitis, enterocolitis, hepatitis, pituitary inflammation, vasculitis myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after normal hormone replacement therapy).

   may be included after normalization of hormone replacement therapy).
4. patients with asthma requiring medical intervention with bronchodilators
5. patients with uncontrolled cardiac clinical symptoms or disease, such as. (1) NYHA class II or higher heart failure. (2) Unstable angina pectoris. (3) Myocardial infarction within 1 year. (4) Clinically significant supraventricular or ventricular arrhythmias requiring clinical (4) patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention.
6. active infection or unexplained fever of >38.5°C (0.5 mg/kg) during screening or before the first dose Fever >38.5°C (in the judgment of the investigator, subjects with fever due to tumor fever can be enrolled).
7. a known history or evidence of interstitial lung disease or active non-infectious pneumonia
8. have a congenital or acquired immune deficiency (e.g., HIV-infected), active Hepatitis B (HBV-DNA ≥ 104 copies/mL) or Hepatitis C (Hepatitis C antibody positive and HCV-RNA above the lower limit of detection for the assay).
9. prior treatment with other PD-1 monoclonal antibodies or other immunotherapy against PD-1/PDL1
10. known hypersensitivity to macromolecular protein agents, or to any of the components of kareolizumab sensitization.
11. Requirement for corticosteroids (>10 mg/day, prednisone) within 14 days prior to first administration of study drug.

10 mg/day, prednisone efficacy dose) or other immunosuppressive agents for systemic therapy within 14 days prior to the first Subjects on systemic therapy with corticosteroids (> 10 mg/day, prednisone efficacy dose) or other immunosuppressive agents within 14 days prior to first study drug administration. In the absence of active autoimmune disease In the absence of active autoimmune disease, inhaled or topical steroids and adrenaline at doses >10 mg/day, prednisone efficacy dose are allowed.

Adrenocorticosteroid replacement at efficacious doses of prednisone. 12. have received an antitumor monoclonal antibody (mAb) within 4 weeks prior to the first administration of study drug (mAb) within 4 weeks prior to the first administration of study drug, or adverse events from previously received drugs have not Recovery (i.e., ≤ grade 1 or at baseline level). Note: Occurrence of ≤ grade 2 neuropathy or ≤ grade 2 alopecia.

Note: Subjects with ≤ grade 2 neuropathy or ≤ grade 2 alopecia are excluded if the subject has undergone major surgery.

If the subject has undergone major surgery, the toxic effects and/or complications of the surgical intervention must be adequately addressed prior to initiation of treatment.

Subjects who have undergone major surgery must have recovered sufficiently from the toxic effects and/or complications of their surgical intervention prior to initiation of treatment.

13. the subject is participating in another clinical study 14. the subject has received a live vaccine within 4 weeks prior to the first administration of the study drug and is allowed to receive injectable 14. Receipt of inactivated viral vaccine for seasonal influenza, by injection, but not receive live attenuated influenza vaccine administered via intranasal route. 15. subjects who, in the judgment of the investigator, have other factors that may force them to terminate the other factors that, in the judgment of the investigator, may force him or her to terminate the study, such as other serious illnesses (including mental illness) requiring comorbid treatment, severely abnormal laboratory test values, family or social factors that circumstances that may affect the safety of the subject or the collection of trial data.

16. other circumstances that, in the judgment of the investigator, make inclusion in this study inappropriate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 3 years
  Objective response rate, according to RECISTv1.1, the proportion of patients with CR or PR was determined. If the patient has not undergone a post-baseline assessment, it is considered unremission.

SECONDARY OUTCOMES:
PFS | up to 3 years
  progression-free survival (PFS) refers to the time from enrollment to the first recording of disease progression as determined by RECISTv1.1, or to death due to any cause (whichever occurs first). PFS will be analyzed in the ITT analysis set.
OS | up to 3 years
  Overall survival (OS) refers to the time from enrollment to the first recorded death due to any cause (whichever occurs first).
HRQoL | up to 3 years
  HRQoL uses EORTCQLQ-C30 to assess the overall health of patients. The post-baseline score of the treatment group was studied, and the score changes from the baseline were summarized descriptively.
HRQoL | up to 3 years
  HRQoL uses EORTCQLQ-OES18 to assess the overall health of patients. The post-baseline score of the treatment group was studied, and the score changes from the baseline were summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Li, doctor, Study Chair — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital & Institute, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No